CLINICAL TRIAL: NCT00335023
Title: Well Being of Obstetric Patients on Minimal Blood Transfusions
Acronym: WOMB
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanquin Research & Blood Bank Divisions (Other)
Collaborators: Erasmus Medical Center (Other)
Responsible Party: Dick van Rhenen, Sanquin Blood Bank South West Region
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01-021b; 0904 (Other Grant/Funding Number: Landsteiner Foundation for Blood Transfusion Research); NTR335 (Registry Identifier: Nederlandse Trial Registratie)
Record Dates: First submitted 2006-06-07; First posted 2006-06-08 (Estimated); Last update posted 2011-07-20 (Estimated); Status verified 2011-07

CONDITIONS: Anemia
Keywords: postpartum hemorrhage; red blood cell transfusion; health related quality of life
MeSH Terms: conditions — Anemia; Postpartum Hemorrhage | interventions — Erythrocyte Transfusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Red blood cell transfusion (Active Comparator): At least one unit of red blood cells will be administered.
  Interventions: Other: Red blood cell transfusion
- Control (No Intervention): No red blood cell transfusion. Iron suppletion is allowed and can be administered according to local protocol. If suppletion is prescribed, the type and duration will be registered

INTERVENTIONS:
Other: Red blood cell transfusion — At least one unit of red blood cells will be administered. The target Hb value after transfusion is at least 8.7 g/dL.
  Arms: Red blood cell transfusion

SUMMARY:
Postpartum haemorrhage (PPH) is one of the top five causes of maternal mortality in developed and developing countries. The most important treatment of PPH is red blood cell (RBC) transfusion. The decision whether to prescribe RBC transfusion is mostly based on postpartum haemoglobin (Hb) values. RBC transfusion should be aimed to reduce morbidity and especially to improve Health Related Quality of Life (HRQoL). The goal of the WOMB study is to assess the effect of RBC transfusion on HRQoL and to confirm the role of HRQoL in deciding whether RBC transfusion is necessary.

DETAILED DESCRIPTION:
The WOMB study is a multicenter trial in patients with PPH, where a restrictive RBC transfusion policy will be compared with a more liberal RBC transfusion policy. Primary outcome in this study is fatigue measured with the MFI questionnaire. Inclusion criteria are: 1) 12-24 h after VD or CS; 2) 4.8 ≤Hb≤ 7.9 g/dL; 3) blood loss ≥ 1000mL or Hb decrease ≥ 1,9 g/dL; 4) age≥ 18 years; 5) no anaemic symptoms. Patients will be randomised for a RBC transfusion or not. The total follow-up period is 6 weeks. HRQoL will be measured at T=0 (12-24 hours postpartum) 3 days, 1, 3 and 6 weeks postpartum. At T=0 and 6 weeks postpartum Hb value will be measured. For the patients who receive a RBC transfusion, the effect of the RBC transfusion will be measured with the Hb value, Hct, platelet and leukocyte count, and the temperature of the patient before and after the RBC transfusion. The sample size is 500 patients: 250 allocated to a RBC transfusion and 250 patients allocated to a restrictive policy.

ELIGIBILITY:
Inclusion Criteria:

* Women older than 18 years
* 12-24 hours after delivery (vaginal or caesarean section)
* Patients are in a clinical obstetric setting
* Blood loss of more than 1000 mL or Hb decrease ≥ 1,9 g/dL
* Hb value between 4.8 g/dL and 7.9 g/dL
* Working knowledge of the national language
* Written consent for participating this study (informed consent)

Exclusion Criteria:

* Patients with severe preeclampsia/ HELLP syndrome
* RBC transfusion during or after delivery but before t=0
* Patients with malignancy
* Patients with severe congenital haemolytic disease, like thalassemia or sickle cell disease
* Patients with compromised immunological status, congenital or acquired by medical treatment or infectious disease (eg. HIV)
* Severe active infectious disease at the time of proposed inclusion
* Severe cardiac, pulmonary, neurological, metabolic or psychiatric co- morbidity (ASA II/III) at the time of proposed inclusion
* Severe physical complaints (tachycardia of more than 100 bpm, dyspnoea, syncope, heart problems) at the time of intended inclusion
* Peripartum death of the newborn, or the newborn being in critical condition on neonatal intensive care

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2004-05; Primary Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Physical Fatigue | on day 3 postpartum
  measured with the MFI questionnaire

SECONDARY OUTCOMES:
Health related quality of life | delivery - six weeks postpartum
  Health related quality of life measured with the following questionnaires: Euro-Qol, SF-36 and the MFI
Blood usage and the costs | delivery - six weeks postpartum
Hemoglobin increase after transfusion | before- after transfusion
  Hb value and platelet count will be measured before and after red blood cell transfusion
Heart beat, blood pressure, temperature | before- after transfusion
  heart beat per minute, blood pressure, temperature will be measured before and after red blood cell transfusion
Hospital stay | delivery - six weeks postpartum
  the hospital stay after delivery will be compared between both arms. All admissions in the first 6 weeks postpartum will be registered
Physical complications (infections, thromboembolic events, hemodynamic events, cardiac events, neurologic events, secondary HPP, obstetric interventions, 'rescue' RBC transfusion) with WHO CTC grade 2 or more. | delivery - six weeks postpartum
  all complications and admissions in the first 6 weeks postpartum will be registered

CONTACTS AND LOCATIONS:
Overall Officials: Dick J van Rhenen, Prof MD PhD, Study Chair — Sanquin Blood Bank South West Region; Johannes J Duvekot, MD, PhD, Study Chair — Department Obstetrics of Erasmus Medical center; Babette W Prick, M.D., Principal Investigator — Department Obstetrics of Erasmus Medical center
Locations (1):
- Sanquin Blood Bank South West Region, Rotterdam, Netherlands

REFERENCES:
- [Derived] Carson JL, Stanworth SJ, Dennis JA, Fergusson DA, Pagano MB, Roubinian NH, Turgeon AF, Valentine S, Trivella M, Doree C, Hebert PC. Transfusion thresholds and other strategies for guiding red blood cell transfusion. Cochrane Database Syst Rev. 2025 Oct 20;10(10):CD002042. doi: 10.1002/14651858.CD002042.pub6. PMID 41114449
- [Derived] Carson JL, Stanworth SJ, Dennis JA, Trivella M, Roubinian N, Fergusson DA, Triulzi D, Doree C, Hebert PC. Transfusion thresholds for guiding red blood cell transfusion. Cochrane Database Syst Rev. 2021 Dec 21;12(12):CD002042. doi: 10.1002/14651858.CD002042.pub5. PMID 34932836
- [Derived] Prick BW, Schuit E, Mignini L, Jansen AJ, van Rhenen DJ, Steegers EA, Mol BW, Duvekot JJ; EBM Connect Collaboration. Prediction of escape red blood cell transfusion in expectantly managed women with acute anaemia after postpartum haemorrhage. BJOG. 2015 Dec;122(13):1789-97. doi: 10.1111/1471-0528.13224. Epub 2015 Jan 20. PMID 25600160
- [Derived] Prick BW, Jansen AJ, Steegers EA, Hop WC, Essink-Bot ML, Uyl-de Groot CA, Akerboom BM, van Alphen M, Bloemenkamp KW, Boers KE, Bremer HA, Kwee A, van Loon AJ, Metz GC, Papatsonis DN, van der Post JA, Porath MM, Rijnders RJ, Roumen FJ, Scheepers HC, Schippers DH, Schuitemaker NW, Stigter RH, Woiski MD, Mol BW, van Rhenen DJ, Duvekot JJ. Transfusion policy after severe postpartum haemorrhage: a randomised non-inferiority trial. BJOG. 2014 Jul;121(8):1005-14. doi: 10.1111/1471-0528.12531. Epub 2014 Jan 10. PMID 24405687
- [Derived] Prick BW, Steegers EA, Jansen AJ, Hop WC, Essink-Bot ML, Peters NC, Uyl-de Groot CA, Papatsonis DN, Akerboom BM, Metz GC, Bremer HA, van Loon AJ, Stigter RH, van der Post JA, van Alphen M, Porath M, Rijnders RJ, Spaanderman ME, Schippers DH, Bloemenkamp KW, Boers KE, Scheepers HC, Roumen FJ, Kwee A, Schuitemaker NW, Mol BW, van Rhenen DJ, Duvekot JJ. Well being of obstetric patients on minimal blood transfusions (WOMB trial). BMC Pregnancy Childbirth. 2010 Dec 16;10:83. doi: 10.1186/1471-2393-10-83. PMID 21162725
- See also: study website — http://www.studies-obsgyn.nl/womb